CLINICAL TRIAL: NCT05693896
Title: Treating Binge Eating and Obesity Digitally in Black Women: A Feasibility Study
Brief Title: Treating Binge Eating and Obesity Digitally in Black Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-2718; 5K23DK129832 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Binge Eating; Binge-Eating Disorder; Weight Gain Prevention; Obesity
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centering Appetite Intervention, Then Attention- Control Group (Experimental): Participants randomized to the attention-control group will participate remotely via a smartphone app and online lessons. The intervention will build participants' self-efficacy to reduce binge eating and to assist them in preventing weight gain.
  Interventions: Behavioral: Centering Appetite
- Attention- Control Group, Then Centering Appetite Intervention (No Intervention): Participants randomized to the centering appetite intervention group will receive weekly psychoeducation emails about general wellness topics, discussion of binge eating, diet, and physical activity.

INTERVENTIONS:
Behavioral: Centering Appetite — A digital treatment of Appetite Awareness Treatment (AAT) and behavioral weight loss treatment (BWL) over 6 months, delivered remotely using Zoom. The goal of AAT is to enable participants to be able to relearn their stomach's hunger signals and begin to obey and monitor functions of satiety. AAT has been successful in helping participants diagnosed with Binge Eating Disorder (BED) and bulimia nervosa reduce binge eating, overeating, urges to eat in response to non-appetite stimuli, and prevent weight gain.
  Arms: Centering Appetite Intervention, Then Attention- Control Group

SUMMARY:
More than 30% of Black women with obesity binge eat. Binge eating may increase the risk for the development of metabolic syndrome and binge-eating-disorder (BED), which is associated with severe obesity. Though several effective treatments for binge eating exist, Black women have not fared well. Not only has their inclusion in treatment trials been limited, but when participating, they are more likely to drop out, and/or lose less weight, compared to their White counterparts. Furthermore, treatment for binge eating is often not available in primary care and community-based settings places where Black women are more likely to receive treatment for their eating and weight-related concerns. Currently, there is scant intervention research to treat binge eating in Black women. With the highest rates of obesity (57%) nationally, Black women are in need of culturally-relevant treatments for binge eating and weight gain prevention. Given the established relationship between frequent binge eating and subsequent weight gain, addressing binge eating among Black women with obesity is imperative.

DETAILED DESCRIPTION:
Aim 1. Modify and adapt a validated program to be a culturally-relevant digital health tool for binge eating and weight management for Black women (BMI > 30 kg/m^2) who binge eat.

Aim 1a. Identify the barriers and facilitators to detecting and treating binge eating in Black women with obesity, and identify strategies for optimizing digital health tools to engage and retain this population.

Aim 1b. Conduct usability testing with a group of stakeholders to guide content and design refinements; refine tool.

Aim 2. In a randomized clinical trial, examine the feasibility and preliminary efficacy of the digital health appetite awareness + behavioral weight program in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* BMI ≥ 30 kg/m^2,
* have and regularly use a Bluetooth-enabled smartphone,
* report at least one binge eating episode weekly,
* work or live within 30 miles of Kannapolis, NC,
* complete the screening questionnaire

Exclusion Criteria:

* currently pregnant,
* in substance abuse treatment,
* involved in another weight reduction program,
* have a history of anorexia,
* are purging,
* currently in treatment for eating difficulties,
* are concurrent intravenous drug users
* consume >4 alcoholic beverages/day

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Recruitment): Total Number of Eligible Adults Enrolled in the Study | 3 month
  Recruitment is defined as the number of potential eligible adults screened for the study versus the number of persons who enrolled in the study.
Retention: Percentage of Participants Retained in the Study | 6 months
  Percentage of eligible participants who were enrolled and retained in the study through the 6 months.
Attendance: Percentage of Intervention Sessions Attended | 6 months
  Percentage of intervention sessions attended for the duration of the study by each participant.

SECONDARY OUTCOMES:
Change from Baseline to Month 3 in weight regain | Baseline, 3 months
  Participant body weight will be measured by trained research staff using calibrated digital scales, with participants in light indoor clothing, with pockets emptied and belts and shoes removed.
Change from Baseline to Month 6 in weight regain | Baseline, 6 months
  Participant body weight will be measured by trained research staff using calibrated digital scales, with participants in light indoor clothing, with pockets emptied and belts and shoes removed.
Change in number of Binge Eating Episodes from Baseline to Month 3 | Baseline, 3 months
  Participant binge eating episodes will be self-monitored via the digital health tool.
Change in number of Binge Eating Episodes from Baseline to Month 6 | Baseline, 6 months
  Participant binge eating episodes will be self-monitored via the digital health tool.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Goode, PhD,MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No